CLINICAL TRIAL: NCT03521999
Title: Randomized Controlled Trial of AboutFace: A Novel Video Storytelling Resource to Improve Access, Engagement, and Utilization of Mental Health Treatment Among Veterans With PTSD
Brief Title: The Use of a Novel Peer Education Program for Improving PTSD Treatment Engagement Among Veterans
Acronym: AboutFace
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IIR 17-123
Record Dates: First submitted 2018-04-26; First posted 2018-05-11 (Actual); Results first posted 2024-06-14 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-01

CONDITIONS: PTSD; Posttraumatic Stress Disorder
Keywords: PTSD; peer resource; Veterans; web-based intervention; digital story telling
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: 376 Veterans who are referred for a PTSD evaluation through the Charleston VAMC PTSD Clinic Team (PCT) and Telehealth Programs and are recommended for PTSD specialty care will be randomized to receive an online peer-to-peer digital storytelling resource [AboutFace] or an educational brochure for PTSD [enhanced Usual Care; eUC]
Who Masked: Outcomes Assessor
Masking Description: Post-treatment assessors and a co-investigator in charge of randomization will be blind to condition assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- AboutFace (Active Comparator): Veterans in the AboutFACe arm will receive access to an online peer-to-peer digital storytelling resource for Veterans with PTSD
  Interventions: Behavioral: AboutFace
- Enhanced Usual Care (eUC) (Placebo Comparator): Veterans in the Enhanced Usual Care (eUC) arm will receive an education brochure for PTSD
  Interventions: Other: Enhanced Usual Care (eUC)

INTERVENTIONS:
Behavioral: AboutFace — AboutFace is an online peer-to-peer digital storytelling resource for Veterans with PTSD. Veterans will have access to AboutFace while they are enrolled in PTSD specialty care through the Charleston PCT.
  Arms: AboutFace
Other: Enhanced Usual Care (eUC) — Enhanced Usual Care (eUC) includes access to a PTSD educational brochure. Veterans will have access to the brochure information while they are enrolled in PTSD specialty care through the Charleston PCT.
  Arms: Enhanced Usual Care (eUC)

SUMMARY:
Behavioral health problems among Veterans have raised awareness of the critical need for more reliable, effective, and accessible ways to recognize those in need, direct them to help, and ensure that they receive the best evidence-based care available. AboutFace is a novel peer education program that features the personal stories of Veterans and is designed to improve Veterans' likelihood of engaging in Post Traumatic Stress Disorder (PTSD) specialty care. Using a randomized controlled study design the investigators propose to compare the efficacy of AboutFace relative to standard care for improving treatment engagement and outcomes. Additional data from VA providers will provide valuable information on wide scale implementation and dissemination of AboutFace. If AboutFace increases access of services, data will have broad implications for overcoming barriers to care for Veterans with PTSD and other stigmatized conditions.

DETAILED DESCRIPTION:
Anticipated Impacts on Veterans Health Care: Behavioral health problems among Veterans have raised awareness of the critical need for more reliable, effective, and accessible means to recognize those in need, direct them to help, and ensure that they receive the best treatment available. Research has suggested that people are most responsive to advice and education when it comes from someone to whom they can relate. AboutFace is a peer education resource for Veterans that was developed, launched, and recently updated by the National Center for PTSD (NCPTSD) based on Health Services Research &Development (HSR&D) funded pilot data. AboutFace features personal stories of Veterans and is designed to improve mental health treatment engagement among Veterans with PTSD and related comorbidities. The study team, which includes the NCPTSD, recently completed a usability assessment and pilot feasibility trial of AboutFace under HSR&D grant #14-360-1. Data from this study (1) guided improvements to AboutFace for increasing PTSD treatment initiation and engagement; and (2) demonstrated the feasibility of the methodology for the proposed study. If AboutFace is found to increase Veterans' initiation and engagement in PTSD treatment, study data will have broad implications for overcoming barriers to care for Veterans with PTSD and other stigmatized conditions.

Background: At least 1 in 10 Veterans meet criteria for PTSD related to their military experience. Treatment for PTSD is widely available, and national dissemination initiatives have increased Veterans' access to best-practice interventions. However, treatment-seeking remains strikingly low; most Veterans with PTSD do not seek mental health services due to perceived stigma and other barriers. NCPTSD developed and launched AboutFace, a public awareness campaign to help Veterans recognize PTSD and motivate them to seek evidence-based care. Since its development, AboutFace has earned three major awards and has had tens of thousands of visits. Despite the tremendous potential for AboutFace to reduce stigma, improve attitudes toward mental health treatment seeking, and to increase PTSD treatment initiation and engagement, it has yet to be formally evaluated or effectively implemented within Veterans Health Administration (VHA) practice settings. In addition to providing needed data on the efficacy of AboutFace and identifying strategies for effective implementation within VHA, this study will provide a greater understanding of the role and value of digital storytelling interventions to improve access to care for a wide range of stigmatized conditions.

Objectives: The primary objectives of the study are to examine the impact of AboutFace on a) increasing PTSD treatment initiation and engagement; and b) decreasing stigma and negative attitudes toward mental health services. It is anticipated that Veterans in the AboutFace condition will be more likely to access and complete treatment than those receiving enhanced Usual Care (eUC) for PTSD. Finally, qualitative interviews with key stakeholders across the nation will be conducted to inform best practices for future implementation of AboutFace.

Methods: A total of 376 Veterans referred for a PTSD assessment and recommended for treatment in the Charleston PTSD clinic will be enrolled in the study. Veterans will be randomized to receive AboutFace versus eUC. All Veterans will receive standard PTSD educational materials, and half will also be randomly assigned to receive AboutFace. Comparisons will be made across indices of treatment engagement [i.e., initiated treatment (yes/no), total number of sessions completed;]; changes in stigma and attitudes toward seeking mental health treatment; and changes in PTSD symptoms and quality of life. Veterans will be assessed on these indices at baseline, 1-month, 3-month, and 6-months.

ELIGIBILITY:
Inclusion Criteria:

* Veterans must be referred for a PTSD evaluation through the Charleston VAMC PTSD Clinic Team (PCT) and Telehealth Programs and recommended for PTSD specialty care through the clinic.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anouk L. Grubaugh, PhD MA BS, Principal Investigator — Ralph H. Johnson VA Medical Center, Charleston, SC
Locations (1):
- Ralph H. Johnson VA Medical Center, Charleston, SC, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bunnell BE, Davidson TM, Hamblen JL, Cook DL, Grubaugh AL, Lozano BE, Tuerk PW, Ruggiero KJ. Protocol for the evaluation of a digital storytelling approach to address stigma and improve readiness to seek services among veterans. Pilot Feasibility Stud. 2017 Feb 17;3:7. doi: 10.1186/s40814-017-0121-3. eCollection 2017. PMID 28239485
- [Result] Hamblen JL, Grubaugh AL, Davidson TM, Borkman AL, Bunnell BE, Ruggiero KJ. An Online Peer Educational Campaign to Reduce Stigma and Improve Help Seeking in Veterans with Posttraumatic Stress Disorder. Telemed J E Health. 2019 Jan;25(1):41-47. doi: 10.1089/tmj.2017.0305. Epub 2018 May 10. PMID 29746232

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Veterans will be referred following a PTSD evaluation through the Charleston VAMC PTSD Clinic Team (PCT) and Telehealth Programs and recommended for PTSD specialty care through the clinic
Period: Completed 1 Month Up
Arm/Group | AboutFace | Enhanced Usual Care (eUC)
Started | 165 | 165
Completed | 106 | 107
Not Completed | 59 | 58
Not completed — Lost to Follow-up | 59 | 58
Period: Completed 3 Month Follow up
Arm/Group | AboutFace | Enhanced Usual Care (eUC)
Started | 165 (Starting N is not based on previous assessment period numbers. If a participant did not complete their 1 month follow up, they are still eligible to complete their 3 and 6 month assessment points.) | 165 (Starting N is not based on previous assessment period numbers. If a participant did not complete their 1 month follow up, they are still eligible to complete their 3 and 6 month assessment points.)
Completed | 101 | 105
Not Completed | 64 | 60
Not completed — Lost to Follow-up | 64 | 59
Not completed — Death | 0 | 1
Period: Completed 6 Month Follow
Arm/Group | AboutFace | Enhanced Usual Care (eUC)
Started | 165 (Starting N is not based on previous assessment period numbers. If a participant did not complete their 1 month follow up, they are still eligible to complete their 3 and 6 month assessment points.) | 164 (Starting N is not based on previous assessment period numbers. If a participant did not complete their 1 month follow up, they are still eligible to complete their 3 and 6 month assessment points. N reduced by one after 1 participant death.)
Completed | 99 | 94
Not Completed | 66 | 70
Not completed — Lost to Follow-up | 66 | 70

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AboutFace | Enhanced Usual Care (eUC) | Total
Number analyzed (Participants) | 165 | 165 | 330
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 157 | 161 | 318
  >=65 years | 8 | 4 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.39 (11.57) | 43.17 (11.78) | 43.78 (11.68)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Missing one data point from Control
  Participants
    number analyzed (Participants) | 165 | 164 | 329
    Female | 57 | 46 | 103
    Male | 108 | 118 | 226
Race (NIH/OMB) [Count of Participants; unit: Participants] — Unknown category captures Hispanic and those who stated "other"
  Participants
    American Indian or Alaska Native | 1 | 1 | 2
    Asian | 2 | 3 | 5
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 76 | 86 | 162
    White | 78 | 68 | 146
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 8 | 7 | 15
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 165 | 165 | 330
Marital Status [Count of Participants; unit: Participants] — Population: One data point missing from Marital status
  Participants
    number analyzed (Participants) | 165 | 164 | 329
    Married | 106 | 104 | 210
    Separated | 6 | 3 | 9
    Divorced | 29 | 29 | 58
    Never Married | 16 | 22 | 38
    Widowed | 2 | 1 | 3
    Other | 6 | 5 | 11
Employment Status [Count of Participants; unit: Participants] — Population: 2 data points missing from Baseline assessment
  Participants
    number analyzed (Participants) | 165 | 163 | 328
    Full Time | 79 | 85 | 164
    Retired | 22 | 18 | 40
    Part Time | 25 | 17 | 42
    Student | 15 | 15 | 30
    Unemployed | 24 | 28 | 52
Combat Veteran status [Count of Participants; unit: Participants] — Population: 3 data points missing for Combat Era
  Participants
    number analyzed (Participants) | 165 | 162 | 327
    No Combat | 48 | 52 | 100
    WWII/Korea | 1 | 1 | 2
    Vietnam | 5 | 2 | 7
    Desert Storm | 17 | 10 | 27
    OEF/OIF | 92 | 93 | 185
    Other | 2 | 4 | 6

OUTCOME MEASURES:

1. Primary Outcome: PTSD Treatment Engagement (Yes/no)
Description: Dichotomous yes/no variable for whether or not a participant started at least one session of PTSD specialty care within 60 days of baseline. This measure indicates the number of participants who attended a minimum of one session of a PTSD treatment within 60 days of the initial baseline administration.
Time Frame: Baseline up to 60 days
Measure: Count of Participants; unit: Participants
Arm/Group | AboutFace | Enhanced Usual Care (eUC)
Number analyzed (Participants) | 165 | 165
Participants | 137 | 132

2. Primary Outcome: Total Number of PTSD Treatment Sessions
Description: Total number of PTSD treatment sessions completed from baseline to 60 days
Time Frame: Baseline up to 60 days
Measure: Mean (Standard Deviation); unit: Number of sessions
Arm/Group | AboutFace | Enhanced Usual Care (eUC)
Number analyzed (Participants) | 165 | 165
Number of sessions | 8.5 (4.8) | 8.5 (4.4)

3. Secondary Outcome: Posttraumatic Stress Disorder Checklist-5 (PCL-5)
Description: The PCL is a 20-item self-report measure of PTSD severity. The self-report rating scale is 0-4 for each symptom: "Not at all," "A little bit," Moderately," "Quite a bit," and "Extremely." Total score can range from 0-80.
Time Frame: 6 months
Population: The overall number of participants analyzed is inconsistent with the total number of participants enrolled in each condition because these results are reflective of the 6 month assessment point. These numbers reflect the number of participants who completed this measure at the 6 month assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AboutFace | Enhanced Usual Care (eUC)
Number analyzed (Participants) | 99 | 91
score on a scale | 49.9 (16.5) | 46.9 (19.7)

4. Secondary Outcome: Endorsed and Anticipated Stigma Inventory (EASI)
Description: EASI assesses different dimensions of stigma-related beliefs about mental health among military personnel and Veterans. It measures 5 dimensions: beliefs about mental illness, beliefs about mental health treatment, beliefs about seeking treatment, concerns about stigma from loved ones, and concerns about stigma in the workplace. Scores range from 40- 200. Higher scores are indicative of greater stigma; thus improvement is evident in reduction of scores/reduction of stigma in mental health.
Time Frame: 6 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AboutFace | Enhanced Usual Care (eUC)
Number analyzed (Participants) | 99 | 91
score on a scale | 99.33 (30.97) | 98.76 (30.45)

5. Secondary Outcome: Patient Health Questionnaire (PHQ-8)
Description: The PHQ-8 is a brief questionnaire that scores each of the 8 Diagnostic Statistical Manual (DSM)-IV criteria for depression as "0" (not at all) to "3" (nearly every day) with higher total scores indicating greater symptoms. Scores range from 0-24. PHQ-8 scores of 5, 10, 15, and 20 represent mild, moderate, moderately severe, and severe depression respectively.
Time Frame: 6 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AboutFace | Enhanced Usual Care (eUC)
Number analyzed (Participants) | 99 | 91
score on a scale | 15.3 (5.7) | 14.5 (6.3)

6. Secondary Outcome: Quality of Life Index (QLI)
Description: The QLI is a 2-part, 33-item self-report measure of life satisfaction and importance regarding various aspects of life with higher scores representing better outcomes. Scores range from 0-30. An increase in score would represent an increase in life satisfaction.
Time Frame: 6 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AboutFace | Enhanced Usual Care (eUC)
Number analyzed (Participants) | 98 | 90
score on a scale | 15.5 (2.6) | 15.5 (2.5)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected throughout entirety of study and reported at time of event. Participant charts were reviewed at each assessment point; 1 month, 3 month and 6 month.
Arm/Group | AboutFace | Enhanced Usual Care (eUC)
All-Cause Mortality (participants affected / at risk) | 0/165 | 1/165
Serious Adverse Events (participants affected / at risk) | 0/165 | 0/165
Other Adverse Events (participants affected / at risk) | 3/165 | 3/165
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AboutFace (N=165) | Enhanced Usual Care (eUC) (N=165)
Inpatient (Psychiatric disorders) | 2 | 3
Incarceration (Social circumstances) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-31): https://cdn.clinicaltrials.gov/large-docs/99/NCT03521999/Prot_SAP_000.pdf